

## Consent Form for Participants Able to Give Consent

Centre name (if applicable): Study Protocol number:

**Full Title of Project:** Frequency of nocturnal hypoglycaemia in adults with insulin treated diabetes and adrenal failure using prednisolone or hydrocortisone: a pilot study (HYPO-DIAD).

Name of Principal Investigator: Dr Monika Reddy

Please initial box

| 1. | I confirm that I have read and understand the participant information sheet version |
|---|---|
| 2. | I understand that my participation is voluntary, and I am free<br>to withdraw at any time, without giving any reason and<br>without my legal rights nor treatment / healthcare being<br>affected. |
| 3. | I agree to my GP being informed of my participation in the study and of any problems that may occur during the study |
| 4. | I understand that sections of any of my medical notes may be looked at by responsible individuals from Imperial College Healthcare NHS Trust or from regulatory authorities where it is relevant to my taking part in this research. |
| 5. | I understand that tissue samples and / or data collected from me are a gift donated to Imperial College Healthcare NHS Trust and that I will not personally benefit financially if this research leads to an invention and/or the successful development of a new test, medication treatment, product or service. |



| <ol> <li>I do/ do not(delete/mark<br/>contacted about the poss<br/>studies.</li> </ol> | as applicable) give conser<br>sibility to take part in other i | <u> </u> |
|---|---|---|
| 7. I understand that the information collected about me will be used to support future research, and may be shared pseudoanonymously with other researchers | | |
| <ol> <li>I understand that pseudo<br/>downloaded from glucose<br/>study</li> </ol> | anonymised data may be<br>e monitoring devices for us | e in the |
| I acknowledge that Dexcom is a separate data controller and is separate from Imperial College Healthcare Trust. | | |
| 10.I agree to receive a written summary of the main findings of this study. (OPTIONAL) | | |
| 11.I consent to take part in "Frequency of nocturnal hypoglycaemia in adults with insulin treated diabetes and adrenal failure using prednisolone or hydrocortisone: a pilot study (HYPO-DIAD).". | | |
| Name of participant | Signature | Date |
| Name of person taking consent | <br>Signature | <br>Date |
| 1 copy for participant; 1 copy | for Principal Investigator 1 | copy for hospital notes |

To ensure confidence in the process and minimise risk of loss, all consent forms must be printed, presented and stored in double sided format

Frequency of nocturnal hypoglycaemia in patients with insulin treated diabetes and adrenal failure using prednisolone or hydrocortisone: a pilot study (HYPO-DIAD). IRAS ID 319768 Consent v1.1 08/03/2023